CLINICAL TRIAL: NCT06371924
Title: Mechanistic Evaluation of Machine Perfusion Strategies in Donation After Circulatory Death Liver Transplantation
Brief Title: Immunometabolism of Machine Perfusion Strategies
Acronym: iMaps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCH23-156
Record Dates: First submitted 2024-02-13; First posted 2024-04-17 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Intervention Model Description: The investigators propose to conduct a randomised clinical trial in which 36 DCD human livers will be allocated to 1 of 3 treatment arms:
  i) SCS; ii)NRP; and iii) HOPE. This will be followed by a period of time in NMP in order to study the IRI response and determine if the quality of the livers is good enough to proceed to transplantation. This study will allow the doctors to decipher the mechanisms of liver IRI in humans in a much better way than what has been achieved to date.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Static Cold Storage (Active Comparator): The donor liver will be flushed in situ with 4C UW preservation solution (or HTK) through the aorta and portal vein, retrieved, and transported to the transplant centre in an icebox.
  Interventions: Device: Machine Perfusion
- Normothermic Regional Perfusion (Active Comparator): The donor aorta and inferior cava vein will be cannulated, followed by descending thoracic aorta cross-clamp and initiation of perfusion (Cardiohelp device) with the donor's own blood at 37C for 2h (while monitoring pump flow, venous O2 saturation, lactate and ALT), followed by in-situ flush with 4C preservation solution as in SCS arm.
  Interventions: Device: Machine Perfusion
- Hypothermic oxygenated perfusion (Active Comparator): The liver will be retrieved and preserved as in SCS arm. Then, on arrival to the transplant unit, the portal vein and hepatic artery will be cannulated, and the liver perfused with hypothermic oxygenated solution (VitaSmart device) for 2h.
  Interventions: Device: Machine Perfusion

INTERVENTIONS:
Device: Machine Perfusion — The quality of DCD organs can be improved by replacing the icebox (static cold storage or SCS), which remains the main approach to preserve the livers after having been retrieved, by strategies that perfuse the livers in a machine (machine perfusion or MP). There are currently 3 MP strategies employed in the clinic: normothermic regional perfusion (NRP) is used in the donors by perfusing the liver with the donor's blood at 37 degrees Celsius, and normothermic (NMP) or hypothermic (HOPE) perfusion are used in the procured livers out of the body (using warm or cold perfusion fluids, respectively). To date, no controlled objective comparisons of these different MP strategies have been undertaken and the doctors do not have a good understanding of their mechanisms of action.

SUMMARY:
There are not enough donated livers for everybody who needs one, and as a result, thousands of patients worldwide are waiting for liver transplants, with many dying while waiting for a life-saving organ. One reason for this shortage is that some usable livers from donors who are considered of high risk are being thrown away out of concern that they might not work well after transplantation due to a problem called ischaemia reperfusion injury (IRI).

The discarded organs are mostly those coming from donors who have died due to cardiac arrest (called 'donation after circulatory death' or DCD), with only 27% of them being used in the UK. The quality of these DCD organs could be improved by changing how they are preserved after being removed from the donor. The most commonly used strategy is still to remove the livers and put them in an icebox ('static cold storage' or SCS). The alternative approaches, which are more complex and expensive, but that can also improve the quality of the DCD livers, involve using machines to pump fluids through the livers ('machine perfusion' or MP).

There are three MP methods being used in patients: 1) normothermic regional perfusion (NRP), which involves pumping the donor's blood through the liver after the donor has died but the liver is still in the donor's body; 2) normothermic machine perfusion (NMP), in which the liver is pumped with blood outside of the donor's body; and 3) hypothermic machine perfusion (HOPE), which is also used outside of the donor's body by pumping cold fluid into the liver. HOPE and NRP have been shown to improve how well DCD livers function after transplantation. NMP can also improve the quality of the DCD livers, but its main advantage is that it allows confirming that the donated liver functions well before proceeding with the transplant. Until now, there has not been a proper comparison of these methods, and the doctors do not understand well the mechanisms through which MP improves the quality of the DCD livers.

The iInvestigators plan to conduct a study where 36 DCD human livers will be split into three groups: SCS, NRP, and HOPE. After that, they will be put in NMP to confirm that they are good enough to be transplanted and to study the mechanisms through which NRP, SCS and HOPE work.

DETAILED DESCRIPTION:
Liver transplant numbers do not meet the existing needs, thousands of patients remain on transplant waiting lists worldwide and many die while awaiting a life-saving organ. A key contributor to organ shortage is the discarding of viable organs coming from donors considered high-risk, for fear that they might malfunction after transplantation as a result of a phenomenon called ischaemia reperfusion injury (IRI). Most of the discarded livers are those donated after circulatory death (DCD), only 27% of which are currently utilised in the UK. The quality of DCD organs can be improved by replacing the icebox (static cold storage or SCS), which remains the main approach to preserve the livers after having been retrieved, by strategies that perfuse the livers in a machine (machine perfusion or MP). There are currently 3 MP strategies employed in the clinic: normothermic regional perfusion (NRP) is used in the donors by perfusing the liver with the donor's blood at 37 degrees Celsius, and normothermic (NMP) or hypothermic (HOPE) perfusion are used in the procured livers out of the body (using warm or cold perfusion fluids, respectively). To date, no controlled objective comparisons of these different MP strategies have been undertaken and doctors do not have a good understanding of their mechanisms of action. The investigators hypothesise that the benefits of MP will depend on the capacity of these strategies to improve the damage to the liver cell mitochondria, which constitutes the first event that elicits IRI at the time of transplantation. To determine this, the investigators propose to conduct a randomised clinical trial in which 36 DCD human livers will be allocated to 1 of 3 treatment arms: i) SCS; ii) NRP; and iii) HOPE. This will be followed by a period of time in NMP in order to study the IRI response and determine if the quality of the livers is good enough to proceed to transplantation. Following transplantation, patients will be followed for up to 12 months.

Our proposal will include three key objectives:

1. To investigate the role of mitochondrial damage in the IRI that takes place when DCD livers are transplanted.
2. To determine the mechanisms through which the different MP strategies influence IRI in DCD liver transplantation.
3. To develop markers to assess the quality of the livers while they are being perfused using NMP before being transplanted into patients.

Our study will allow us to decipher the mechanisms of liver IRI in humans in a much better way than what has been achieved to date. Furthermore, it will provide guidelines as to the best way of employing the MP technologies and may result in the identification of new treatments. Ultimately, our proposal will serve to improve the quality of DCD livers and increase the number of patients who can safely receive a liver transplant.

ELIGIBILITY:
Inclusion Criteria Donor inclusion criteria

1. DCD category III donors considered for abdominal organs-only retrieval.
2. Donor age ≥18 years.
3. Retrieval procedure allocated to KCH or UHB NORS teams.
4. Donor liver accepted for a patient at KCH or UHB transplant waiting list via the standard offering process.
5. Functional donor warm ischaemia (defined as a period between the systolic blood pressure <50mmHg and aortic cold flush) ≤30 minutes.
6. Donor BMI <35kg/m2.
7. Predicted cold ischaemic time <8 hours.
8. Donor family has given consent to use donated liver for research.

Transplant recipient inclusion criteria

1. Recipients 18 years of age or older.
2. Listed on an elective transplant waiting list.
3. First liver transplantation.
4. Suitable to receive a DCD graft based on the liver listing MDT.
5. Willingness to consent for the study participation.

Exclusion Criteria Donor exclusion criteria

1. Donor is HIV, hepatitis B (HBV HbsAg) or hepatitis C (HCV RNA) positive. HBV anti-Hbc positive donors are acceptable.
2. Macroscopic evidence of fibrosis.
3. Liver weight >2.5 kg.
4. Retrieval of cardiothoracic organs intended for transplantation.
5. Any medical condition that, in the opinion of the principal investigator, would interfere with safe completion of the trial.

Transplant recipient exclusion criteria

1. High-risk surgical candidates (i.e. presence of extensive portomesenteric thrombosis, previous complex upper abdominal surgery).
2. Patients receiving super-urgent transplantation for acute and acute-on-chronic liver failure.
3. Patients unable to give full informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of different preservation strategies on the development of mitochondrial damage following reperfusion during NMP. | 2 years
  changes in mitochondrial complex I enzyme activity in liver tissue samples obtained 30 minutes and 4 hours after initiating NMP, as assessed by an established spectrophotometric assay (values will be reported as a ratio to citrate synthase)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No